CLINICAL TRIAL: NCT01629771
Title: Disability and Quality of Life in Patients With Lymphatic Filariasis in Rural Southern India
Status: Completed | Type: Observational
Sponsor: Northwestern University (Other)
Responsible Party: Principal Investigator, Roopal Kundu, Assistant Professor of Dermatology, Northwestern University
Other Study IDs: STU63944
Record Dates: First submitted 2012-06-26; First posted 2012-06-28 (Estimated); Results first posted 2013-08-02 (Estimated); Last update posted 2014-03-20 (Estimated); Status verified 2014-02

CONDITIONS: Lymphatic Filariasis
MeSH Terms: conditions — Elephantiasis, Filarial

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Lymphatic Filariasis
- Patients without Lymphatic Filariasis

SUMMARY:
According to the World Health Organization, lymphatic filariasis, a mosquito-borne parasitic disease, is the second leading cause of disability worldwide. Across 81 countries, approximately 120 million people are infected with the disease, and of those infected, an estimated 40% reside in India alone. The most disfiguring symptoms of lymphatic filariasis, elephantiasis and lymphedema, cause long-term suffering in patients who are then often embarrassed or even rejected from their communities. Because of the disease's debilitating physical and social effects on patients, this study will explore the intersection of disability and health-related quality of life (HRQoL) in lymphatic filariasis patients in India. Specifically, HRQoL and disability in lymphatic filariasis subjects and age- and gender- matched control subjects will be compared. Two HRQoL tools , the general Dermatology Life Quality Index (DLQI) and a disease-specific instrument developed by a dermatology group in India will be used to gauge HRQol. In addition, the demographic and disease-specific factors associated with HRQoL and disability in filarial lymphedema subjects will be identified.

ELIGIBILITY:
Case Inclusion Criteria

* Subjects with a clinical diagnosis of lymphatic filariasis
* Subjects over the age of 18 and able to give consent

Case Exclusion Criteria

* Subjects on active treatment for lymphatic filariasis
* Subjects who are under the age of 18 or unable to give informed consent

Control Inclusion Criteria

* Subjects without a clinical diagnosis of lymphatic filariasis
* Subjects over the age of 18 and able to give consent

Control Exclusion Criteria

* Subjects without a clinical diagnosis of lymphatic filariasis
* Subjects who are under the age of 18 or unable to give informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: This study will be conducted in the Kasaragod district of Kerala, India. Subjects with a clinical diagnosis of lymphatic filariasis of a single body part or more will be recruited from the Institute of Applied Dermatology, and age-matched controls
Sampling Method: Probability Sample
Enrollment: 72 (Actual)
Dates: Start 2012-05; Primary Completion 2012-06 (Actual); Study Completion 2012-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Roopal Kundu, MD, Principal Investigator — Northwestern University
Locations (2):
- Northwestern University Department of Dermatology, Chicago, Illinois, United States
- Institute of Applied Dermatology, Kasaragod District, Kerala, India

REFERENCES:
- [Background] Michael E, Bundy DA, Grenfell BT. Re-assessing the global prevalence and distribution of lymphatic filariasis. Parasitology. 1996 Apr;112 ( Pt 4):409-28. doi: 10.1017/s0031182000066646. PMID 8935952
- [Background] Coreil J, Mayard G, Louis-Charles J, Addiss D. Filarial elephantiasis among Haitian women: social context and behavioural factors in treatment. Trop Med Int Health. 1998 Jun;3(6):467-73. doi: 10.1046/j.1365-3156.1998.00238.x. PMID 9657509
- [Background] Recommendations of the International Task Force for Disease Eradication. MMWR Recomm Rep. 1993 Dec 31;42(RR-16):1-38. PMID 8145708
- [Background] Dreyer G, Noroes J, Figueredo-Silva J. New insights into the natural history and pathology of bancroftian filariasis: implications for clinical management and filariasis control programmes. Trans R Soc Trop Med Hyg. 2000 Nov-Dec;94(6):594-6. doi: 10.1016/s0035-9203(00)90200-1. No abstract available. PMID 11198637
- [Background] Raju K, Jambulingam P, Sabesan S, Vanamail P. Lymphatic filariasis in India: epidemiology and control measures. J Postgrad Med. 2010 Jul-Sep;56(3):232-8. doi: 10.4103/0022-3859.68650. PMID 20739779
- [Background] Narahari SR, Aggithaya MG, Prasanna KS, Bose KS. An integrative treatment for lower limb lymphedema (elephantiasis). J Altern Complement Med. 2010 Feb;16(2):145-9. doi: 10.1089/acm.2008.0546. No abstract available. PMID 20180687
- [Background] Finlay AY, Khan GK. Dermatology Life Quality Index (DLQI)--a simple practical measure for routine clinical use. Clin Exp Dermatol. 1994 May;19(3):210-6. doi: 10.1111/j.1365-2230.1994.tb01167.x. PMID 8033378
- [Background] International Society of Lymphology. The diagnosis and treatment of peripheral lymphedema. 2009 Concensus Document of the International Society of Lymphology. Lymphology. 2009 Jun;42(2):51-60. No abstract available. PMID 19725269
- See also: Northwestern University Department of Dermatology Actively Enrolling Research Trials — http://www.feinberg.northwestern.edu/depts/dermatology/research/clinical-trials/ctu-active%20trials.htm

RESULTS

PARTICIPANT FLOW:
Groups:
- Subjects With Lymphatic Filariasis: Subjects with lymphatic filariasis completed health-related quality of life questionnaires.
- Control Subjects: Age- and gender-matched control subjects completed health-related quality of life questionnaires.
Period: Overall Study
Arm/Group | Subjects With Lymphatic Filariasis | Control Subjects
Started | 36 | 36
Completed | 36 | 36
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Subjects With Lymphatic Filariasis | Control Subjects | Total
Number analyzed (Participants) | 36 | 36 | 72
Age, Continuous [Mean (Standard Deviation); unit: years] | 51.7 (16.2) | 52.3 (16.1) | 52.0 (16.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 28 | 28 | 56
  Male | 8 | 8 | 16
Region of Enrollment [Number; unit: participants]
  India | 36 | 36 | 72

OUTCOME MEASURES:

1. Primary Outcome: Dermatology Life Quality Index (DLQI) Domain Scores
Description: The DLQI is a 10-item questionnaire measuring skin-specific quality of life through six domains: Symptoms & Feelings, Daily Activities, Leisure, Work & School, Personal Relationships, and Treatment. Symptoms & Feelings, Daily Activities, Leisure, and Personal Relationships are each scored from 0 to 3, where 0 is associated with no effect on a patient's life, and 3 is associated with a large effect on a patient's life. Work & School and Treatment are each scored from 0 to 3, where 0 is associated with no effect on a patient's life, and 6 is associated with a large effect on a patient's life.
Time Frame: Assessed after enrollment
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Subjects With Lymphatic Filariasis | Control Subjects
Number analyzed (Participants) | 36 | 36
units on a scale
  Symptoms & Feelings | 3 [2 to 4] | 0 [0 to 0]
  Daily Activities | 1 [0 to 2] | 0 [0 to 0]
  Leisure | 1 [1 to 3] | 0 [0 to 0]
  Work & School | 0 [0 to 1] | 0 [0 to 0]
  Personal Relationships | 0 [0 to 1] | 0 [0 to 0]
  Treatment | 0 [0 to 1] | 0 [0 to 0]

2. Primary Outcome: Lymphatic Filariasis-Specific Quality of Life (LFSQQ) Domain Scores
Description: The LFSQQ was developed to assess quality of life in subjects with lymphatic filariasis through seven domains: Mobility, Self-Care, Usual Activities, Disease Burden, Pain/Discomfort, Psychological Health, and Social Participation. Items are scored on a 5-point scale (no problem, mild, moderate, severe, most severe), and scores for each domain are calculated based on the number of questions answered and the raw scores. Scores for each domain range from 0 to 100, where 0 is associated with a worse quality of life and 100 is associated with a better quality of life.
Time Frame: Assessed after enrollment
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Subjects With Lymphatic Filariasis | Control Subjects
Number analyzed (Participants) | 36 | 36
units on a scale
  Mobility | 67 [58 to 80] | 100 [88 to 100]
  Self-Care | 100 [82 to 100] | 100 [100 to 100]
  Usual Activities | 92 [75 to 100] | 100 [100 to 100]
  Disease Burden | 63 [60 to 75] | 100 [100 to 100]
  Pain/Discomfort | 90 [83 to 96] | 100 [98 to 100]
  Psychological Health | 75 [64 to 86] | 100 [95 to 100]
  Social Participation | 67 [50 to 85] | 100 [100 to 100]

3. Primary Outcome: World Health Organization Disability Assessment Schedule 2.0 (WHODAS 2.0) Domain Scores
Description: The WHODAS 2.0 is a generic health and disability assessment tool that describes effects of disease on six domains: Cognition, Mobility, Self-Care, Getting Along, Life Activities, and Participation in Society. Responses are measured on a 5-point scale from 1 (no difficulty) to 5 (extreme difficulty or cannot do). Scores are calculated using a WHO SPSS 36 version syntax for employed subjects and a WHO SPSS 32 version syntax for unemployed subjects. Scores for each domain range from 0 to 100, where 0 is associated with no impairment of health status, and 100 is associated with a greater impairment of health status.
Time Frame: Assessed after enrollment
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Subjects With Lymphatic Filariasis | Control Subjects
Number analyzed (Participants) | 36 | 36
units on a scale
  Cognition | 15 [3 to 20] | 0 [0 to 3]
  Mobility | 50 [19 to 69] | 0 [0 to 13]
  Self-Care | 5 [0 to 10] | 0 [0 to 0]
  Getting Along | 25 [0 to 33] | 0 [0 to 0]
  Life Activities | 20 [0 to 40] | 0 [0 to 5]
  Participation in Society | 25 [17 to 38] | 0 [0 to 8]

ADVERSE EVENTS:
Arm/Group | Subjects With Lymphatic Filariasis | Control Subjects
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes